CLINICAL TRIAL: NCT05040399
Title: Sternal Wound Infection in Patients Undergone Sternal Fixation Using Locking Compression Plates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kareem Ahmed Hosny, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AssiutUnivMed
Record Dates: First submitted 2021-08-21; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Sternal Fracture; Sternal Wound Infection; Surgical Site Infection
Keywords: sternum; wound infection; locking compression plates; sternal wires
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Intervention Model Description: Case-Control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Locking Compression Plates (Other): Patients in whom we used Locking compression plates for sternal fixation
  Interventions: Other: Locking Compression Plates
- Wires (Other): Patients in whom we used Sternal Wires for sternal fixation
  Interventions: Other: Sternal Wires

INTERVENTIONS:
Other: Locking Compression Plates — Plates and screws for sternal fixation
  Arms: Locking Compression Plates
Other: Sternal Wires — sternal wires used for fixation of sternum
  Arms: Wires

SUMMARY:
Sternal Wound Infection (SWI) in open heart surgery is one of the most annoying and avoidable complications that one encounters during work. Investigators investigate the rates of sternal wound infection (SWI) in patients in whom were used locking compression plates (LCP) versus in patients in whom were used wires to fixate the sternum for variable causes. SWI increases the overall cost and burden in the medical service and increases the patients suffering and disability. investigators aim to provide our patients with the most suitable means for sternal fixation.

ELIGIBILITY:
Inclusion Criteria:

* All genders are accepted
* Ages from 18 to 80 years old
* Patients undergoing Open heart surgery for any reasons and trauma patients who suffer sternal fractures of any type.

Exclusion Criteria:

* Ages less than 18 years old and older than 80 years old
* Patients undergoing minimally invasive surgeries utilizing access sites other than the sternum.
* Trauma patients with multiple complex injuries.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-20 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Sternal Wound Infection rate | 3 weeks post-operative
  sternal wound infection in the form of redness, hotness, swelling and discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty Of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes